CLINICAL TRIAL: NCT05439694
Title: The Effect of Using Tranexamic Acid Soaked Absorbable Gelatin Sponge in Reducing Rectus Sheath Hematoma Formation After Cesarean Section in Patients Using Warfarin Compounds
Brief Title: TXA Soaked Gelatin Sponge to Reduce Rectus Sheath Hematoma After C.S. in Patients Using Warfarin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Hany, MD, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AymanMscPPH
Record Dates: First submitted 2022-06-22; First posted 2022-06-30 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Rectus Sheath Hematoma; Cesarean Section
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gelatin Sponges soaked with TXA (Experimental): 21 patients will have 2 pieces of Gelatin Sponges (SURGISPON®; AEGIS LIFESCIENCES, India) (Size, 40 cm2) soaked in Tranexamic acid (Kapron, Amoun Pharmaceuticals SAE, Egypt. 5ml Amp, 100mg /1ml) each sponge will be soaked with one ampoule and applied between the anterior rectus sheath and the rectus abdominis muscle, one sponge on each muscle.
  Interventions: Drug: Tranexamic acid
- Gelatin Sponges (Experimental): 2 Gelatin Sponges (SURGISPON®; AEGIS LIFESCIENCES, India) (Size, 40 cm2)
  Interventions: Drug: Tranexamic acid
- NO SPONGE (No Intervention): 21 patients will have no sponge inserted 10 ml of saline

INTERVENTIONS:
Drug: Tranexamic acid — have 2 pieces of Gelatin Sponges (SURGISPON®; AEGIS LIFESCIENCES, India) (Size, 40 cm2) soaked in Tranexamic acid (Kapron, Amoun Pharmaceuticals SAE, Egypt. 5ml Amp, 100mg /1ml)
  Other Names: Gelatin Sponges (SURGISPON®; AEGIS LIFESCIENCES, India)
  Arms: Gelatin Sponges; Gelatin Sponges soaked with TXA

SUMMARY:
The aim of this randomized controlled study is to demonstrate the effect of Local application of TXA impregnated in a gelatin sponge in reducing Rectus sheath hematoma formation in patients treated with warfarin following cesarean section.

DETAILED DESCRIPTION:
The study will include (63) pregnant women attending for cesarean delivery who will receive anticoagulation (warfarin) postnatally.

Patients included in this study will be subjected to:

- Informed consent: patients representing the study population will be counselled about the intervention and informed written consent will be taken.

Consenting patients will be subjected to the following:

1. Detailed personal, obstetric and medical and surgical history. 2- Examination: General Examination.

* Vital signs: Blood pressure, pulse and temperature.
* Weight, height, BMI.
* Abdominal examination for assessment of fundal level. 3. Laboratory Investigations Preoperatively
* CBC, Coagulation Profile, Blood Chemistry. 5. Abdominal Ultrasound: in order to assess the following: a. Gestational age determination. c. Placental site. CS will be done by Senior Obstetricians, Using Standard CS technique, with visceral and parietal peritoneum re-approximation and insertion of a passive intraperitoneal drain. Fascial closure will be done using continuous slowly absorbable sutures. Meticulous hemostasis will be achieved using monopolar cauterization. An active drain (Hemovac®) will be applied in the space between anterior rectus sheath and the rectus abdominis muscle in all patients.

Patients will be randomly assigned into three groups Randomization is done by computer generated random numbers in opaque envelops.

Group 1:

(21) patients will have 2 pieces of Gelatin Sponges (SURGISPON®; AEGIS LIFESCIENCES, India) (Size, 40 cm2) soaked in Tranexamic acid (Kapron, Amoun Pharmaceuticals SAE, Egypt. 5ml Amp, 100mg /1ml) each sponge will be soaked with one ampoule and applied between the anterior rectus sheath and the rectus abdominis muscle, one sponge on each muscle.

Group 2:

(21) patients will have 2 Gelatin Sponges (SURGISPON®; AEGIS LIFESCIENCES, India) (Size, 40 cm2) Not impregnated with Tranexamic acid applied locally using the same method as the previous group.

Group 3:

(21) patients will have Neither Gelatin Sponge nor Tranexamic acid applied. Follow up patients for vital signs and manifestations of allergic reactions in the immediate post operative period.

The intraperitoneal drain will be removed after 24 hours in all groups. While the (Hemovac®) drain will be removed after achieving target INR in all groups.

All Patients will be receiving bridging anticoagulation using LMWH(Enoxaparin) alone for 3 days in therapeutic doses (1mg/kg twice daily) to be initiated 12 hours after Surgery in most cases.Then Warfarin will be added on post operative day 3. LMWH will be withdrawn after achieving target INR.

Then comparison between the three groups regarding

* Hemovac® Drain output in cc per day till achieving Target INR Levels for all patients.
* Ultrasound assessment of rectus sheath hematoma if present after achieving Target INR Levels for all patients.

ELIGIBILITY:
Inclusion Criteria:

* o Pregnant women attending for elective CS.

  * Women on antenatal anticoagulation ( LMWH , UFH , Fondaparinux ) for conditions such as : Prosthetic Valve , DVT , Pulmonary embolism , Dural sinus thrombosis , AF.
  * Pregnant Women with indication for postnatal warfarin anticoagulation( Prosthetic Valve , DVT , Dural Sinus Thrombosis , AF , Pulmonary embolism )
  * Age between 20-40 years.
  * Pregnancies between 37 and 39 weeks
  * BMI between (18.5 - 30.0)

Exclusion Criteria:

* o Pregnancy with risk of obstetric hemorrhage such as abnormally invasive placenta, placenta previa, placental abruption.

  * Women with Renal and Hepatic failure
  * Women with bleeding diathesis for reasons other than warfarin anticoagulation therapy
  * Women with known allergy to Tranexamic acid
  * Anemia Hb below 8g/dl

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Rectus sheath hematoma formation | 1 weeks
  Rectus sheath hematoma formation detected by Ultrasound
Excessive bleeding from subrectus space | 1 week
  amount of blood coming out of the drains

SECONDARY OUTCOMES:
Thromboembolic manifestations | 1 weeks
  DVT
Blood transfusion | 1 week
  ml
The need for surgical evacuation of rectus sheath hematoma | 1 week
  surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibbons L, Belizan JM, Lauer JA, Betran AP, Merialdi M, Althabe F. Inequities in the use of cesarean section deliveries in the world. Am J Obstet Gynecol. 2012 Apr;206(4):331.e1-19. doi: 10.1016/j.ajog.2012.02.026. Epub 2012 Mar 1. PMID 22464076
- [Background] Hatjipetrou A, Anyfantakis D, Kastanakis M. Rectus sheath hematoma: a review of the literature. Int J Surg. 2015 Jan;13:267-271. doi: 10.1016/j.ijsu.2014.12.015. Epub 2014 Dec 19. PMID 25529279
- [Background] Cherry WB, Mueller PS. Rectus sheath hematoma: review of 126 cases at a single institution. Medicine (Baltimore). 2006 Mar;85(2):105-110. doi: 10.1097/01.md.0000216818.13067.5a. PMID 16609349
- [Background] Jafferbhoy SF, Rustum Q, Shiwani MH. Abdominal compartment syndrome--a fatal complication from a rectus sheath haematoma. BMJ Case Rep. 2012 Apr 2;2012:bcr1220115332. doi: 10.1136/bcr.12.2011.5332. PMID 22602838
- [Background] Osinbowale O, Bartholomew JR. Rectus sheath hematoma. Vasc Med. 2008 Nov;13(4):275-9. doi: 10.1177/1358863X08094767. PMID 18940904
- [Background] McCormack PL. Tranexamic acid: a review of its use in the treatment of hyperfibrinolysis. Drugs. 2012 Mar 26;72(5):585-617. doi: 10.2165/11209070-000000000-00000. PMID 22397329
- [Background] Liang J, Liu H, Huang X, Xiong W, Zhao H, Chua S, Li Z. Using tranexamic acid soaked absorbable gelatin sponge following complex posterior lumbar spine surgery: A randomized control trial. Clin Neurol Neurosurg. 2016 Aug;147:110-4. doi: 10.1016/j.clineuro.2016.06.001. Epub 2016 Jun 13. PMID 27343711
- [Derived] Hany A, Mansour A, Sediek M, Nabil M. Role of tranexamic acid-soaked gelatin sponge in minimizing rectus sheath hematoma after cesarean section in women treated with warfarin, a simple tool for high-risk cases, a randomized controlled trial. Eur J Med Res. 2023 Oct 20;28(1):448. doi: 10.1186/s40001-023-01434-7. PMID 37864195